CLINICAL TRIAL: NCT05275946
Title: Phase I Investigator-initiated Clinical Trial in Patients With Differentiated Thyroid Cancer (Papillary Cancer, Follicular Cancer) by the Targeted Alpha Therapy Drug TAH-1005 ([211At] NaAt) (Alpha-T1 Study)
Brief Title: Targeted Alpha Therapy Using Astatine (At-211) Against Differentiated Thyroid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Osaka University (Other)
Responsible Party: Principal Investigator, Tadashi Watabe, Assistant Professor, Osaka University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT1-001
Record Dates: First submitted 2022-01-22; First posted 2022-03-11 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Cancer
Keywords: Targeted alpha therapy; Astatine (At-211)
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Other)
  Interventions: Drug: Targeted alpha therapy

INTERVENTIONS:
Drug: Targeted alpha therapy — Single intravenous administration

SUMMARY:
Single intravenous administration of TAH-1005 is performed in patients with differentiated thyroid cancer (papillary cancer, follicular cancer) who cannot obtain therapeutic effect with standard treatment or who have difficulty in implementing and continuing standard treatment. The safety, pharmacokinetics, absorbed dose, and efficacy will be evaluated to determine the recommended dose for Phase II clinical trial.

DETAILED DESCRIPTION:
Radioactive iodine (I-131) has long been used clinically for patients with metastatic differentiated thyroid cancer. However, some patients are refractory to repetitive I-131 treatment, despite the targeted regions showing sufficient iodine uptake. In such patients, beta-particle therapy using I-131 is inadequate and another strategy is needed using more effective radionuclide targeting the sodium/iodide symporter (NIS). Astatine (At-211) is receiving increasing attention as an alpha-emitter for targeted radionuclide therapy. At-211 is a halogen element with similar chemical properties to iodine. Alpha particles emitted from At-211 has higher linear energy transfer as compared to beta particles from I-131 and exert a better therapeutic effect by inducing DNA double strand breaks and free radical formation. Thus, targeted alpha therapy using At-211 is highly promising for the treatment of advanced differentiated thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with differentiated thyroid cancer (papillary cancer, follicular cancer) after total thyroidectomy who meet the following conditions (1) resistance to standard treatment or (2) difficulty in continuing standard treatment (1) Patients who are refractory to standard treatment such as 131I-NaI treatment Insufficient therapeutic effect after 3 or more 131I-NaI treatments. 131I-NaI treatment resistance and difficulty in performing or continuing tyrosine kinase inhibitor (TKI) treatment (2) Patients who have difficulty continuing standard treatment such as 131I-NaI treatment Ablation for residual thyroid or 131I-NaI treatment for relapsed / metastatic lesions has been performed, but relapsed / metastatic lesions were observed at the time of participation in this study, and 131I-NaI is the standard treatment. If it is difficult to continue treatment or if local radiation therapy (including addition) is not indicated (if it is not 131I-NaI treatment resistant, TKI treatment is not indicated).
2. Patients aged 18 years or older at the time of consent acquisition
3. Patients with stable general condition with PS (Performance status) of 0 to 2 in ECOG (Eastern Cooperative Oncology Group)
4. Patients who can be expected to survive for 6 months or more, judging from clinical symptoms and medical examination findings
5. Patients with no or controlled brain metastases with symptoms
6. Patients with no clinically significant abnormal findings in electrocardiogram, respiratory rate, and blood oxygen saturation within 30 days before registration
7. Patients whose laboratory values within 30days before the enrollment are within the range specified in the protocol
8. Patients who thoroughly listened to the explanation of the clinical trial, agreed to the examination, visit during the observation period and follow-up survey, contraception during the clinical trial period, etc. according to the clinical trial protocol, and signed the consent document.

Exclusion Criteria:

1. Patients who need fertility preservation
2. Pregnant or potentially pregnant women, lactating patients
3. Patients with active double cancer (simultaneous double cancer and ectopic double cancer with a disease-free period of 5 years or less)
4. Patients who received other investigational or unapproved drugs within 5 weeks prior to enrollment
5. Patients who received chemotherapy, immunotherapy or radiation therapy within 8 weeks prior to enrollment in this study
6. Patients with uncontrollable active infections
7. HBsAg positive, HCV antibody positive or HIV antibody positive patients
8. Patients with mental illness or psychiatric symptoms who are judged to be difficult to participate in clinical trials
9. Other patients who are judged to be inappropriate by the investigator, etc.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse events as assessed by CTCAE v5.0 | From the start of iodine restriction to 6 months after administration
  Type, severity, frequency of occurrence and duration of adverse events
Dose Limiting Toxicity | within 4 weeks after administration
  Toxicity is defined as one or more of the following items for which a causal relationship with the investigational drug cannot be ruled out.
  1. Grade 3 * hematological toxicity that lasts for 7 days or more
  2. Hematological toxicity of Grade 4 * or higher regardless of duration
  3. Febrile neutropenia regardless of duration
  4. Thrombocytopenia with bleeding tendency or requiring platelet transfusion
  5. Anemia requiring red blood cell transfusion
  6. Neutropenia with infection
  7. Non-hematological toxicity of Grade 3 * or higher that does not improve with symptomatic treatment and lasts for 7 days or longer. However, the following are excluded.
     * Abnormal laboratory test values that are not clinically significant
     * Toxicity that can be controlled to Grade 2 * or less with maximum supportive care
     * Due to exacerbation of the underlying disease (*: Grade specified in CTCAE v.5.0J COG version)

SECONDARY OUTCOMES:
Blood pressure | within 4 weeks after administration
  Systolic and diastolic blood pressure (mmHg)
Heart rate | within 4 weeks after administration
  Pulse (bpm)
Blood oxygen saturation | within 4 weeks after administration
  Percutaneous oxygen saturation (%)
Respiratory rate | within 4 weeks after administration
  Respiratory rate (times/min)
Body temperature | within 4 weeks after administration
  Body temperature (°C)
Body weight | within 4 weeks after administration
  Weight (kg)
Symptoms and examination findings | within 4 weeks after administration
  Subjective symptoms and medical examination findings
Hematological examination | within 4 weeks after administration
  White blood cell count (/μL), red blood cell count (×10^4/μL), hemoglobin (g/dL), hematocrit (%), platelet count (×10^4/μL)
Blood biochemical test | within 4 weeks after administration
  Total protein (g/dL), albumin (g/dL), total bilirubin (mg/dL), AST (U/L), ALT (U/L), ALP (U/L), γ-GTP (U/L), LDH (U/L), total cholesterol (mg/dL), triglyceride (mg/dL), uric acid (mg/dL), BUN (mg/dL), creatinine (mg/dL), CK (U/L), Na (mmol/L), K (mmol/L), Cl (mmol/L), Ca (mmol/L), CRP (mg/dL)
Urinalysis | within 4 weeks after administration
  Urinary protein, urine sugar, urineous blood, urobilinogen (qualitative test)
12-lead ECG | within 4 weeks after administration
  Presence or absence of abnormal findings in waveform
Pharmacokinetic parameters 1) | until 24 hours after administration
  AUC (Area under the plasma concentration versus time curve, Bq·min/mL)
Pharmacokinetic parameters 2) | until 24 hours after administration
  AUC / D (Area under the plasma concentration versus time curve divided by injected dose, min/mL)
Pharmacokinetic parameters 3) | until 24 hours after administration
  Cmax (Peak plasma concentration, Bq/mL)
Pharmacokinetic parameters 4) | until 24 hours after administration
  Cmax / D (Peak plasma concentration divided by injected dose, /mL)
Pharmacokinetic parameters 5) | until 24 hours after administration
  Tmax (Time to maximum plasma concentration, min)
Pharmacokinetic parameters 6) | until 24 hours after administration
  T1 / 2 (Time from Tmax to half of maximum plasma concentration, min)
Pharmacokinetic parameters 7) | until 24 hours after administration
  CL (Clearance, L/hr/kg)
Pharmacokinetic parameters 8) | until 24 hours after administration
  Vss (Volume of distribution in steady state, L/kg)
Excretion 1) urinary | until 24 hours after administration
  Urine volume (mL) and radioactivity (Bq): Radioactivity and volume will be combined to report radioactivity concentration (Bq/mL).
Excretion 2) fecal | until 24 hours after administration
  Stool weight (g) and radioactivity (Bq): Radioactivity and weight will be combined to report radioactivity concentration (Bq/g).
Excretion 3) exhaled | until 24 hours after administration
  Exhaled volume (mL) and radioactivity (Bq): Radioactivity and volume will be combined to report radioactivity concentration (Bq/mL).
Radioactivity concentration in major organs | until 24 hours after administration
  Changes in radioactivity concentration (Bq/mL) in major organs over time: Whole-body imaging (planar and SPECT/CT) is performed to evaluate the distribution in the body at 1 hour, 3 hours, 24 hours after the administration.
Residence time of major organs | until 24 hours after administration
  Residence time (hr) of each organ
Absorbed dose of major organs | until 24 hours after administration
  Absorbed dose (mGy / MBq) of each organ
Preliminary effectiveness assessment 1) | 3 and 6 months after administration
  Evaluation of treatment effect on CT images by referring to the Revised RECIST guideline (version 1.1): CR (Complete response), PR (Partial response), SD (Stable disease), or PD (Progressive disease)
Preliminary effectiveness assessment 2) | 3 and 6 months after administration
  Evaluation of uptake change in diagnostic [131I] NaI scans: CR , PR, SD, or PD
Preliminary effectiveness assessment 3) | 3 and 6 months after administration
  Evaluation of changes in tumor markers: blood thyroglobulin (ng/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka University Hospital, Suita, Japan

IPD SHARING:
Plan to Share IPD: Undecided